CLINICAL TRIAL: NCT01821053
Title: Urine-plasminogen as a Predictor for Development Of Preeclampsia in Pregnant Women With Type 1 Diabetes Mellitus
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Lise Hald Nielsen, doctor, Ph.D student, Odense University Hospital
Other Study IDs: 1-10-72-1-13
Record Dates: First submitted 2013-03-26; First posted 2013-03-29 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Preeclampsia; Type 1 Diabetes
Keywords: Preeclampsia; Pregestational Type 1 diabetes; diabetes mellitus; proteinuria; plasminogen; plasmin; renin; aldosterone; angiotensin; epithelial sodium channel; ENaC
MeSH Terms: conditions — Pre-Eclampsia; Diabetes Mellitus, Type 1; Diabetes Mellitus; Proteinuria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood serum plasma urine
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pregestational type 1 diabetes: It is an observational study. No intervention is made.

SUMMARY:
A tonic active epithelial Na+ channel (ENaC) in pre-eclampsia (PE) escaped normal hormonal control may offer an attractive explanatory model for the pathophysiology of established PE. The channel is activated by plasmin. Microalbuminuria predicts the development of pre-eclampsia in pregnant patients with pregestational diabetes type 1. The investigators hypothesize that urine-plasmin excreted in the kidneys, when proteinuria occurs, could be the cause. The investigators want to test the correlation between measurable plasmin/plasminogen in the urine early in pregnancy and the development of preeclampsia in pregnant patients with type 1 diabetes.

DETAILED DESCRIPTION:
Study aim and hypothesis:

Aim:

To test whether there is a measurable correlation between plasmin/plasminogen, abnormally excreted in the kidneys, and the development of pre-eclampsia in pregnant women with Type 1 diabetes.

Hypothesis:

1. The amount of proteases ( plasmin/plasminogen ), excreted in urine, predicts development of preeclampsia in pregnant patients with type 1 diabetes.

If a correlation between excreted plasmin/plasminogen, in urine, in patients with type 1 diabetes and development of preeclampsia, are seen, proteases might be used as a marker for pre-eclampsia in this group of patients. Prospectively perhaps also as a marker for disease severity.

In these high risk groups it is possible that outpatient visits could be optimized and thus lower the amount of preterm births.

Study design:

The study is an observational, longitudinal - prospective study. Women with pregestational type 1 diabetes are included when they show up for their first outpatient pregnancy visit around pregnancy week 9.

Selection of patients:

Patients are selected from Gynecological- obstetric department, Aarhus University hospital - Skejby, and Gynecological- Obstetric department, Odense University Hospital. To be included they must be singleton-pregnant, have turned 18 years and have Type 1 diabetes.

Background information:

Date of birth, sex, weight, height, BMI, smoking status, current medical treatment, duration of diabetes and parity are registered.

Length of gestation, placental weight, way of delivery (natural birth or cesarean section), umbilical cord pH, apgar score and infant weight are registered post-partum.

Effect variables:

Clinical:

Weight, height, BMI, smoking status, microalbuminuria/proteinuria. Blood pressure (systolic, diastolic, mean arterial pressure). Weight of placenta.

Blood test measurements:

Se-creatinine, p-Na+, p-K+. P-plasminogen, P-albumin, Aldosterone.

Measurements in 50 ml "spot urine":

Plasmin, plasminogen, ENaC peptide fragment (analyses in location of development,) Proteolytic activity, Prostatin, Creatinine, Na+, K+, Aldosterone, Albumin

Study process:

Collection of blood- and spot-urine samples:

Urine-samples are collected in pregnancy week 9-14. Blood pressure is measured. Samples and blood-pressures are re-collected in pregnancy-week 20, 28,32, 36 and perhaps 38.

Following outcomes are observed: Development of preeclampsia, defined by hypertension ( > 140/90 mmHg), and proteinuria ( >0,3 g/24 hour). Preterm delivery and light for gestational age.

Data- analysis methods:

This is an observational longitudinal-prospective study which includes approximately 130 pregnant patients with Type 1 diabetes. Patients are included from Skejby and Odense University Hospitals in cooperation.

Results are evaluated statistically by uni - and multivariate logistic regression analysis.

Population size estimation:

Similar (Danish) observational prospective studies on urine- biomarkers (including albumin) ability to predict preeclampsia/preterm delivery, in patients with pre-gestational type 1 diabetes, have been made. They achieved high significance data with spot-samples of 130 -170 patients. With the participation of two centers it seems realistic and adequately to include 130 patients within the settings of a Ph. D. study. Every year an amount of 50-60 patients are seen in the outpatient ward at Skejby- and Odense University Hospitals (in all approximately 100-120 patients).

ELIGIBILITY:
Inclusion Criteria:

* singleton gravida,
* over 18 years,
* Pregestational type 1 diabetes. Gestation week 8-14.

Exclusion Criteria:

1. Possible comorbidity like systemic lupus erythematosus (SLE), hypertension and rheumatoid arthritis.
2. Organic or systematic diseases with clinical relevance ( ex. Malignity)

However it has to be mentioned that quite some patients have thyroid diseases with no impact on the kidneys nor hypertension. It is therefore possible to include these patients.

Thyroid diseases are NOT a reason for exclusion.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: pregnant women with pregestational type 1 diabtes are included when they show up for their first outpatient pregnancy visit around the 9th weeks gestation.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2013-06; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
preeclampsia | 3 years
  The development of preeclampsia, defined by hypertension ( > 140/90 mmHg) and proteinuria ( >0,3 g/24 hour).

SECONDARY OUTCOMES:
preterm delivery | 3 years
  post-partum registration of preterm delivery
light for gestational age | 3 years
  post-partum registration of "light for gestational age"

CONTACTS AND LOCATIONS:
Overall Officials: Boye L. Jensen, Professor, Study Director — cardiovascular and renal research department, Odense University Hospital
Locations (1):
- Gynelogical Obstetrical Department, Skejby, Aarhus N, Denmark

REFERENCES:
- [Derived] Isaksson GL, Nielsen LH, Palarasah Y, Jensen DM, Andersen LLT, Madsen K, Bistrup C, Jorgensen JS, Ovesen PG, Jensen BL. Urine excretion of C3dg and sC5b-9 coincide with proteinuria and development of preeclampsia in pregnant women with type-1 diabetes. J Hypertens. 2023 Feb 1;41(2):223-232. doi: 10.1097/HJH.0000000000003288. PMID 36583350
- [Derived] Nielsen LH, Jensen BL, Fuglsang J, Andersen LLT, Jensen DM, Jorgensen JS, Kitlen G, Ovesen P. Urine albumin is a superior predictor of preeclampsia compared to urine plasminogen in type I diabetes patients. J Am Soc Hypertens. 2018 Feb;12(2):97-107. doi: 10.1016/j.jash.2017.12.003. Epub 2017 Dec 13. PMID 29305116
- See also: webpage of the research group and related projects — http://www.hupp.dk